CLINICAL TRIAL: NCT01581879
Title: Randomized, 2-way Crossover, Bioequivalence Study of Ziprasidone HCL Capsules, 20 mg in Healthy Subjects Under Fed Conditions.
Brief Title: Bioequivalence Study of Ziprasidone HCL Capsules, 20 mg of Dr. Reddy's Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 40350
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Ziprasidone hydrochloride; crossover
MeSH Terms: interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone HCL Capsules, 20 mg (Experimental): Ziprasidone HCL Capsules, 20 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ziprasidone Hydrochloride
- Geodon Capsules, 20 mg (Experimental): Geodon Capsules, 20 mg of Pfizer Inc
  Interventions: Drug: Ziprasidone Hydrochloride

INTERVENTIONS:
Drug: Ziprasidone Hydrochloride — Ziprasidone HCL Capsules, 20 mg
  Other Names: Geodon

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of ziprasidone 20 mg capsules versus Geodon 20 mg capsules under fed conditions.

DETAILED DESCRIPTION:
Randomized, 2-way crossover, bioequivalence study of Ziprasidone 20 mg capsules and Geodon 20 mg capsules in healthy subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, smoker or non-smoker, 18 years of age and older.
* Capable of consent.
* BMI between 19.0 and 30.0 kg/m2 inclusively.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 100 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or heart rate less than 60 or over 100 bpm) at screening.
* Qtc > 430 for males and Qtc > 450 for females.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit ( more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reaction to heparin, ziprasidone, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazole, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms(e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological endocrinal cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptives.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows.

  1. 50 mL to 300 mL of whole blood within 30 days,
  2. 301 mL to 500 mL of whole blood within 45 days, or
  3. more than 500 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* History or known presence of tardive dyskinesia.
* History of neuroleptic malignant syndrome.
* History or known presence of clinically significant cardiac diseases (such as heart failure, QT prolongation, congenital long QT syndrome, myocardial infarction, cardiac arrhythmias, conduction abnormalities) or other conditions such as electrolyte disturbance, hypokalemia or hypomagnesemia.
* Breast-feeding subject.
* Positive urine pregnancy test at screening.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-steril male partner (i.e male who has not been sterilized by vasectomy for at least 6 months ) within 14 days prior to study drug administration. Acceptable methods of contraception.

  1. intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration;
  2. condom or diaphragm + spermicide;
  3. hormonal contraceptives (starting at least 4 weeks prior to study drug administration.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | 1, 2, 3, 3.50, 4, 4.50, 5, 5.50, 6, 6.50, 7, 8, 9, 10, 12, 16, 24 and 36 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R. Pizarro, MD, Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC Ft. Myers, Inc., Fort Myers, Florida, United States